CLINICAL TRIAL: NCT04976101
Title: A Pilot Study to Assess Sinusoidal Galvanic Vestibular Stimulation in Neurogenic Orthostatic Hypotension
Brief Title: Sinusoidal Galvanic Vestibular Stimulation for Neurogenic Orthostatic Hypotension / Syncope
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It never enrolled any patients
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro2020-0755
Record Dates: First submitted 2021-07-09; First posted 2021-07-26 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Neurogenic Orthostatic Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinusoidal Galvanic Vestibular Stimulation (Experimental): Treatment:
  1. Stimulation of the vestibular nerves with 0.025 Hz, 2 mA sinusoidal galvanic vestibular stimulation Depending on initial results, changes in frequency may range up to 0.1 Hz.
  Interventions: Device: Sinosuidal Galvanic Vestibular Stimulation
- Placebo (Placebo Comparator): Treatment:
  1. Placebo (sham) (no current given however the electrodes and devise is placed and computer keys pressed). Depending on initial results, changes in frequency may range up to 0.1 Hz.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Sinosuidal Galvanic Vestibular Stimulation — stimulus will be given by applying paste electrodes over the mastoid processes and plugging the leads into a battery driven-stimulus box, which when activated by a switch, will provide a very low frequency (VLF) bipolar, ± 2 mA, 0.025 Hz oscillating current sGVS between the mastoids
  Arms: Sinusoidal Galvanic Vestibular Stimulation
Device: Placebo — When assigned to placebo arm of the study, the patients will undergo same procedure as the treatment, only current will not be passed. (the device will still be placed on the mastoid process)
  Arms: Placebo

SUMMARY:
Neurogenic orthostatic hypotension occurs in a significant number of people and has no effective treatment. Neurogenic orthostatic hypotension is associated with intermittent episodes of fainting which can be debilitating for the patients. Using sinusoidal galvanic vestibular stimulation, an oscillating current between the two ears, collaborators have discovered an effective technique to habituate anesthetized rats that develop vasovagal responses. The investigators propose to determine whether a similar use of sinusoidal galvanic vestibular stimulation can eliminate or alleviate neurogenic orthostatic hypotension and the associated syncope in susceptible human subjects. If so, then sinusoidal galvanic vestibular stimulation, which is safe and widely used to study muscle sympathetic nerve activity, can be used in humans, who have a history of syncope and a positive tilt test to habituate vasovagal responses. Habituation will be accomplished using repetitive periods of sinusoidal galvanic vestibular stimulation in two 30min sessions three times/week for 2 weeks. Similar 1 hour sessions are routinely used by others when activating muscle sympathetic nerve activity with sinusoidal galvanic vestibular stimulation without harm to the subjects. The 30 min periods were chosen because this was effective in producing habituation of vasovagal responses. The habituating stimulus will be given by applying paste electrodes over the mastoid processes and plugging the leads into a battery driven-stimulus box, which when activated by a switch, will provide a very low frequency bipolar, ± 2 mA, 0.025 Hz oscillating current sinusoidal galvanic vestibular stimulation between the mastoids. Subjects will be seated during the stimulation. The onset and end of the stimulation period will be denoted by tones, and the subjects will be free to watch television, read, or listen to music while they are being stimulated. The effectiveness of the habituation will be determined in several ways: 1) Subjects will keep a history of the number of episodes of syncope in the inter-test intervals. 2) They will have tilt tests at the beginning and end of habituation. 3) Their blood pressure and heart rate will be recorded and the investigators will determine if there is a loss of low frequency (0.025 Hz) oscillations, which the investigators have found in animal models to disappear when the animals are habituated. 4) Habituation should be accompanied by an increase in heart rate to counteract the fall in blood pressure.

DETAILED DESCRIPTION:
Syncope is a highly prevalent condition affecting 42% of the population at some point in life. Physical injury occurs with syncopal events and the danger of injury becomes more prevalent with age. Syncope accounts for 3% of visits to emergency departments and 6% of all admissions to hospitals. For patients with frequent recurrent syncope, psychosocial impairment has an estimated adverse impact on 33% of the assessed aspects of daily life. There is also a large economic impact, with an estimated $2.4 billion annual cost, mostly due to hospitalizations.

Neurogenic orthostatic hypotension (nOH) results from impaired arterial vasoconstriction that normally is mediated by the baroreflex in response to gravitational pooling of blood. The characteristic findings in nOH are a drop in systolic blood pressure (SBP) of 20 mmHg or more, or a drop in diastolic blood pressure (DBP) of 10 mmHg or more, in response to standing or head-up tilt. What distinguishes nOH from other causes of orthostatic hypotension, such as vasovagal syncope or dehydration, is a blunted compensatory heart rate increase (<15 BPM). nOH accounts for 15% of syncope in the general population and 24% of such cases in emergency room setting. The autonomic failure that precipitates nOH may result from α-synuclein protein deposits in central glial cells (multiple system atrophy) or in postganglionic autonomic neurons when associated with Parkinson's disease or primary autonomic failure. Secondary causes of autonomic failure include diabetic neuropathy and other autoimmune conditions that selectively target the peripheral autonomic nerves.

There is currently no standard of care for people suffering from syncope. Several treatment options have been explored, including beta blockers, corticosteroids, and pacemakers, but none of these have been more effective than placebo. The most promising therapy to date has been repeated static head-up tilts. Vestibulo-sympathetic reflex (VSR) is a term used for the redistribution of blood by vestibular stimulation through the actions of the sympathetic nervous system. 60° static head-up tilt activates otolith and body tilt receptors, which produce cardiovascular changes through the VSR. Using repeated static head-up tilts, "syncope-sensitive" patients were repetitively tilted 60° for periods of time. This was shown to habituate the (VSR) and reduce or eliminate syncope in some cases. However, while it was possible to habituate some subjects with head-tilts, the habituation techniques were too tedious and impractical to be effective in the general population. If there were a less tedious procedure that activated the vestibular system, it could be used to habituate syncope through the VSR.

Sinusoidal galvanic vestibular stimulation (sGVS) activates the otolith system. Blood pressure (BP) and heart rate (HR) have been studied in vasovagal responses in isoflurane-anesthetized Long-Evans rats during sinusoidal galvanic vestibular stimulation (sGVS) and nose-up tilt. In these studies, susceptible rats developed synchronous ≈20-50 mmHg decreases in BP and ≈20-50 bpm decreases in HR over seconds that recovered slowly over minutes in response to repeated vestibular (otolith) stimulation. The sudden decrease in BP and HR, followed by the slower return to pre-stimulus values, are the main components of the vasovagal response that underlie and generate vasovagal syncope. It was found that rats previously susceptible to the induction of vasovagal responses progressively lost their susceptibility as testing continued. The loss of susceptibility to vasovagal responses indicates that the rats were habituated through activation of the VSR, using sGVS. It was concluded that habituation was successful by blocking the occurrence of low frequency oscillations in BP and HR in rats, which are thought to be the critical elements in initiating vasovagal responses. The loss of susceptibility in this study was associated with a rise in HR to oppose the fall in BP. These findings concurred with previous studies demonstrating habituated responses with static head-up tilts. Why these findings were not supported by some other studies, remains unclear; but one author suggested the reason for their findings in humans was that static head-up tilts were sufficiently tedious that it resulted in non-compliance.

The strategy for addressing nOH should likely focus on raising BP rather than HR as a fall in BP is the defining feature of this condition. Studies of the VSR have been performed in rats without identified vasovagal responses. Yakushin and colleagues applied linear acceleration in anesthetized rats and found increases in BP that were maximal during upward and forward translation [36]. HR was unaffected by single translations, but oscillations may influence it more gradually.

There are challenges in the study of various populations affected by syncope. The most common condition, vasovagal syncope may be difficult to objectively diagnose due to the intermittent nature of the symptoms. In particular, many patients have normal tilt testing in the laboratory setting and are only symptomatic during times of physical or emotional stress. A more easily diagnosed condition, postural orthostatic tachycardia syndrome, is far less common and patients frequently improve spontaneously after adolescence.

This study will focus on syncope caused by nOH because there is a larger population of potential subjects and laboratory testing is more reliable. It is our hypothesis that sinusoidal galvanic vestibular stimulation (sGVS) can be used to produce habituation of syncope in humans. sGVS has been used to activate muscle sympathetic nerve activity (MSNA) without side-effects beyond motion-sickness in a few test subjects. During habituation periods, subjects are able to read, listen to music, and watch TV, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unexpected intermittent syncope or a positive tilt test

Exclusion Criteria:

* Syncope cannot be related to significant heart disease
* cannot be not be related to serious medical illnesses that cause increased susceptibility to fainting, such as in Parkinson's Disease
* Pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Net change in blood pressure during head-up tilt | 1 week prior vs 1 week after treatment
  Blood pressure is measured during a head up tilt test and recorded
Net change in heart rate during head-up tilt | 1 week prior vs 1 week after treatment
  Heart rate is measured during a head up tilt test and recorded

SECONDARY OUTCOMES:
Gain of baroreceptor sensitivity | 1 week prior vs 1 week after treatment
  Gain of baroreceptor sensitivity
Phase of baroreceptor sensitivity | 1 week prior vs 1 week after treatment
  Phase of baroreceptor sensitivity
Change in frequency of syncope in the week prior vs week after treatment | 1 week prior vs 1 week after treatment
  Measuring change in frequency of syncope in the week prior vs week after treatment
Change in frequency of low frequency oscillations in blood pressure and heart rate during tilt testing | 1 week prior vs 1 week after treatment
  Measuring the change in frequency of low frequency oscillations in blood pressure and heart rate during tilt testing

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gizzi, MD, Principal Investigator — HUMC NSI
Locations (1):
- Hackensack Univeristy Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] da Silva RM. Syncope: epidemiology, etiology, and prognosis. Front Physiol. 2014 Dec 8;5:471. doi: 10.3389/fphys.2014.00471. eCollection 2014. PMID 25538626
- [Background] Task Force for the Diagnosis and Management of Syncope; European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Heart Failure Association (HFA); Heart Rhythm Society (HRS); Moya A, Sutton R, Ammirati F, Blanc JJ, Brignole M, Dahm JB, Deharo JC, Gajek J, Gjesdal K, Krahn A, Massin M, Pepi M, Pezawas T, Ruiz Granell R, Sarasin F, Ungar A, van Dijk JG, Walma EP, Wieling W. Guidelines for the diagnosis and management of syncope (version 2009). Eur Heart J. 2009 Nov;30(21):2631-71. doi: 10.1093/eurheartj/ehp298. Epub 2009 Aug 27. No abstract available. PMID 19713422
- [Background] Grubb BP. Clinical practice. Neurocardiogenic syncope. N Engl J Med. 2005 Mar 10;352(10):1004-10. doi: 10.1056/NEJMcp042601. No abstract available. PMID 15758011
- [Background] Sun BC. Quality-of-life, health service use, and costs associated with syncope. Prog Cardiovasc Dis. 2013 Jan-Feb;55(4):370-5. doi: 10.1016/j.pcad.2012.10.009. PMID 23472773
- [Background] Arnold AC, Ng J, Lei L, Raj SR. Autonomic Dysfunction in Cardiology: Pathophysiology, Investigation, and Management. Can J Cardiol. 2017 Dec;33(12):1524-1534. doi: 10.1016/j.cjca.2017.09.008. Epub 2017 Sep 14. PMID 29102451
- [Background] Sarasin FP, Louis-Simonet M, Carballo D, Slama S, Junod AF, Unger PF. Prevalence of orthostatic hypotension among patients presenting with syncope in the ED. Am J Emerg Med. 2002 Oct;20(6):497-501. doi: 10.1053/ajem.2002.34964. PMID 12369019
- [Background] Calkins H. Pharmacologic approaches to therapy for vasovagal syncope. Am J Cardiol. 1999 Oct 21;84(8A):20Q-25Q. doi: 10.1016/s0002-9149(99)00626-8. PMID 10568557
- [Background] Cohen B, Martinelli GP, Xiang Y, Raphan T, Yakushin SB. Vestibular Activation Habituates the Vasovagal Response in the Rat. Front Neurol. 2017 Mar 15;8:83. doi: 10.3389/fneur.2017.00083. eCollection 2017. PMID 28360882
- [Background] Sheldon R, Connolly S; Vasovagal Pacemaker Study II. Second Vasovagal Pacemaker Study (VPS II): rationale, design, results, and implications for practice and future clinical trials. Card Electrophysiol Rev. 2003 Dec;7(4):411-5. doi: 10.1023/B:CEPR.0000023157.37745.76. PMID 15071266
- [Background] Yates BJ, Bolton PS, Macefield VG. Vestibulo-sympathetic responses. Compr Physiol. 2014 Apr;4(2):851-87. doi: 10.1002/cphy.c130041. PMID 24715571
- [Background] Yates BJ, Holmes MJ, Jian BJ. Adaptive plasticity in vestibular influences on cardiovascular control. Brain Res Bull. 2000 Sep 1;53(1):3-9. doi: 10.1016/s0361-9230(00)00302-6. PMID 11033202
- [Background] Mittelstaedt H. Origin and processing of postural information. Neurosci Biobehav Rev. 1998 Jul;22(4):473-8. doi: 10.1016/s0149-7634(97)00032-8. PMID 9595557
- [Background] Mittelstaedt H. Somatic graviception. Biol Psychol. 1996 Jan 5;42(1-2):53-74. doi: 10.1016/0301-0511(95)05146-5. PMID 8770370
- [Background] Yates BJ, Miller AD. Properties of sympathetic reflexes elicited by natural vestibular stimulation: implications for cardiovascular control. J Neurophysiol. 1994 Jun;71(6):2087-92. doi: 10.1152/jn.1994.71.6.2087. PMID 7931504
- [Background] Cohen B, Yakushin SB, Holstein GR. What does galvanic vestibular stimulation actually activate: response. Front Neurol. 2012 Oct 22;3:148. doi: 10.3389/fneur.2012.00148. eCollection 2012. No abstract available. PMID 23093948
- [Background] Holstein GR, Friedrich VL Jr, Martinelli GP, Ogorodnikov D, Yakushin SB, Cohen B. Fos expression in neurons of the rat vestibulo-autonomic pathway activated by sinusoidal galvanic vestibular stimulation. Front Neurol. 2012 Feb 28;3:4. doi: 10.3389/fneur.2012.00004. eCollection 2012. PMID 22403566
- [Background] Holstein GR, Friedrich VL Jr, Martinelli GP. Projection neurons of the vestibulo-sympathetic reflex pathway. J Comp Neurol. 2014 Jun 15;522(9):2053-74. doi: 10.1002/cne.23517. PMID 24323841
- [Background] Ector H, Reybrouck T, Heidbuchel H, Gewillig M, Van de Werf F. Tilt training: a new treatment for recurrent neurocardiogenic syncope and severe orthostatic intolerance. Pacing Clin Electrophysiol. 1998 Jan;21(1 Pt 2):193-6. doi: 10.1111/j.1540-8159.1998.tb01087.x. PMID 9474671
- [Background] Ector H. Neurocardiogenic, vasovagal syncope. Eur Heart J. 1999 Dec;20(23):1686-7. doi: 10.1053/euhj.1999.1827. No abstract available. PMID 10562472
- [Background] Foglia-Manzillo G, Giada F, Gaggioli G, Bartoletti A, Lolli G, Dinelli M, Del Rosso A, Santarone M, Raviele A, Brignole M. Efficacy of tilt training in the treatment of neurally mediated syncope. A randomized study. Europace. 2004 May;6(3):199-204. doi: 10.1016/j.eupc.2004.01.002. PMID 15121070
- [Background] Raphan T, Cohen B, Xiang Y, Yakushin SB. A Model of Blood Pressure, Heart Rate, and Vaso-Vagal Responses Produced by Vestibulo-Sympathetic Activation. Front Neurosci. 2016 Mar 31;10:96. doi: 10.3389/fnins.2016.00096. eCollection 2016. PMID 27065779
- [Background] Julu PO, Cooper VL, Hansen S, Hainsworth R. Cardiovascular regulation in the period preceding vasovagal syncope in conscious humans. J Physiol. 2003 May 15;549(Pt 1):299-311. doi: 10.1113/jphysiol.2002.036715. Epub 2003 Apr 4. PMID 12679368
- [Background] Lewis T. A Lecture on VASOVAGAL SYNCOPE AND THE CAROTID SINUS MECHANISM. Br Med J. 1932 May 14;1(3723):873-6. doi: 10.1136/bmj.1.3723.873. No abstract available. PMID 20776843
- [Background] Thomson HL, Wright K, Frenneaux M. Baroreflex sensitivity in patients with vasovagal syncope. Circulation. 1997 Jan 21;95(2):395-400. doi: 10.1161/01.cir.95.2.395. PMID 9008455
- [Background] Kaufmann H, Hainsworth R. Why do we faint? Muscle Nerve. 2001 Aug;24(8):981-3. doi: 10.1002/mus.1102. No abstract available. PMID 11439373
- [Background] Cohen B, Dai M, Ogorodnikov D, Laurens J, Raphan T, Muller P, Athanasios A, Edmaier J, Grossenbacher T, Stadtmuller K, Brugger U, Hauser G, Straumann D. Motion sickness on tilting trains. FASEB J. 2011 Nov;25(11):3765-74. doi: 10.1096/fj.11-184887. Epub 2011 Jul 25. PMID 21788449
- [Background] Yakushin SB, Martinelli GP, Raphan T, Xiang Y, Holstein GR, Cohen B. Vasovagal oscillations and vasovagal responses produced by the vestibulo-sympathetic reflex in the rat. Front Neurol. 2014 Apr 4;5:37. doi: 10.3389/fneur.2014.00037. eCollection 2014. PMID 24772102
- [Background] Cohen B, Martinelli GP, Raphan T, Schaffner A, Xiang Y, Holstein GR, Yakushin SB. The vasovagal response of the rat: its relation to the vestibulosympathetic reflex and to Mayer waves. FASEB J. 2013 Jul;27(7):2564-72. doi: 10.1096/fj.12-226381. Epub 2013 Mar 15. PMID 23504712
- [Background] Nowak JA, Ocon A, Taneja I, Medow MS, Stewart JM. Multiresolution wavelet analysis of time-dependent physiological responses in syncopal youths. Am J Physiol Heart Circ Physiol. 2009 Jan;296(1):H171-9. doi: 10.1152/ajpheart.00963.2008. Epub 2008 Nov 7. PMID 18996985
- [Background] Reybrouck T, Heidbuchel H, Van De Werf F, Ector H. Long-term follow-up results of tilt training therapy in patients with recurrent neurocardiogenic syncope. Pacing Clin Electrophysiol. 2002 Oct;25(10):1441-6. doi: 10.1046/j.1460-9592.2002.01441.x. PMID 12418741
- [Background] Kinay O, Yazici M, Nazli C, Acar G, Gedikli O, Altinbas A, Kahraman H, Dogan A, Ozaydin M, Tuzun N, Ergene O. Tilt training for recurrent neurocardiogenic syncope: effectiveness, patient compliance, and scheduling the frequency of training sessions. Jpn Heart J. 2004 Sep;45(5):833-43. doi: 10.1536/jhj.45.833. PMID 15557724
- [Background] Di Girolamo E, Di Iorio C, Leonzio L, Sabatini P, Barsotti A. Usefulness of a tilt training program for the prevention of refractory neurocardiogenic syncope in adolescents: A controlled study. Circulation. 1999 Oct 26;100(17):1798-801. doi: 10.1161/01.cir.100.17.1798. PMID 10534467
- [Background] Yates BJ, Jian BJ, Cotter LA, Cass SP. Responses of vestibular nucleus neurons to tilt following chronic bilateral removal of vestibular inputs. Exp Brain Res. 2000 Jan;130(2):151-8. doi: 10.1007/s002219900238. PMID 10672468
- [Background] Duygu H, Zoghi M, Turk U, Akyuz S, Ozerkan F, Akilli A, Erturk U, Onder R, Akin M. The role of tilt training in preventing recurrent syncope in patients with vasovagal syncope: a prospective and randomized study. Pacing Clin Electrophysiol. 2008 May;31(5):592-6. doi: 10.1111/j.1540-8159.2008.01046.x. PMID 18439174
- [Background] Yakushin SB, Martinelli GP, Raphan T, Cohen B. The response of the vestibulosympathetic reflex to linear acceleration in the rat. J Neurophysiol. 2016 Dec 1;116(6):2752-2764. doi: 10.1152/jn.00217.2016. Epub 2016 Sep 28. PMID 27683882
- [Background] Gendelman HE, Linzer M, Gabelman M, Smoller S, Scheuer J. Syncope in a general hospital patient population. Usefulness of the radionuclide brain scan, electroencephalogram, and 24-hour Holter monitor. N Y State J Med. 1983 Oct-Nov;83(11-12):1161-5. No abstract available. PMID 6580561
- [Background] Soteriades ES, Evans JC, Larson MG, Chen MH, Chen L, Benjamin EJ, Levy D. Incidence and prognosis of syncope. N Engl J Med. 2002 Sep 19;347(12):878-85. doi: 10.1056/NEJMoa012407. PMID 12239256
- [Background] Klingberg D, Hammam E, Macefield VG. Motion sickness is associated with an increase in vestibular modulation of skin but not muscle sympathetic nerve activity. Exp Brain Res. 2015 Aug;233(8):2433-40. doi: 10.1007/s00221-015-4313-x. Epub 2015 May 30. PMID 26025612
- [Background] Bent LR, Bolton PS, Macefield VG. Modulation of muscle sympathetic bursts by sinusoidal galvanic vestibular stimulation in human subjects. Exp Brain Res. 2006 Oct;174(4):701-11. doi: 10.1007/s00221-006-0515-6. Epub 2006 May 24. PMID 16721608
- [Background] Grewal T, James C, Macefield VG. Frequency-dependent modulation of muscle sympathetic nerve activity by sinusoidal galvanic vestibular stimulation in human subjects. Exp Brain Res. 2009 Aug;197(4):379-86. doi: 10.1007/s00221-009-1926-y. Epub 2009 Jul 7. PMID 19582437
- [Background] Hammam E, James C, Dawood T, Macefield VG. Low-frequency sinusoidal galvanic stimulation of the left and right vestibular nerves reveals two peaks of modulation in muscle sympathetic nerve activity. Exp Brain Res. 2011 Sep;213(4):507-14. doi: 10.1007/s00221-011-2800-2. Epub 2011 Jul 29. PMID 21800255
- [Background] Hammam E, Dawood T, Macefield VG. Low-frequency galvanic vestibular stimulation evokes two peaks of modulation in skin sympathetic nerve activity. Exp Brain Res. 2012 Jun;219(4):441-6. doi: 10.1007/s00221-012-3090-z. Epub 2012 Apr 17. PMID 22526950
- [Background] El Sayed K, Dawood T, Hammam E, Macefield VG. Evidence from bilateral recordings of sympathetic nerve activity for lateralisation of vestibular contributions to cardiovascular control. Exp Brain Res. 2012 Sep;221(4):427-36. doi: 10.1007/s00221-012-3185-6. Epub 2012 Jul 19. PMID 22811217